CLINICAL TRIAL: NCT04354727
Title: Phase Ib/II Study of APG-1252 in Patients With Myelofibrosis Who Progressed After Initial Therapy
Brief Title: A Study of APG-1252 in Patients With Myelofibrosis Who Progressed After Initial Therapy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG1252MU101
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Myelofibrosis
Keywords: JAK2 wild type; JAK2V617F mutation; Thrombocythemia; Polycythemia vera
MeSH Terms: conditions — Primary Myelofibrosis; Thrombocytosis; Polycythemia Vera | interventions — pelcitoclax; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APG-1252 (Experimental)
  Interventions: Drug: APG-1252
- APG-1252 + Ruxolitinib (Experimental)
  Interventions: Drug: APG-1252; Drug: Ruxolitinib

INTERVENTIONS:
Drug: APG-1252 — infusion once weekly
Drug: Ruxolitinib — taken orally twice a day
  Other Names: Jakafi
  Arms: APG-1252 + Ruxolitinib

SUMMARY:
The study is a designed to evaluate safety and activity of APG-1252 when administered as monotherapy and in combination with ruxolitinib in previously ruxolitinib treated myelofibrosis patients.

DETAILED DESCRIPTION:
Part 1 will evaluate safety of APG-1252 monotherapy using a 3+3 dose escalation study design. The starting dose of APG-1252 monotherapy will be 160 mg administered as an intravenous injection over 30 minutes once weekly in a 28-day cycle. If the APG-1252 at 160 mg is tolerated (0/3 and ≤ 1/6 DLTs), dose escalation to 240 mg will be evaluated and declared as recommended phase 2 dose (RP2D) if tolerated. No doses higher than 240 mg once per week will be explored. If the 160 mg once weekly dose schedule is not tolerated (≥ 2/3 or ≥ 2/6 DLTs) de-escalation to 80 mg once weekly dose will be explored. No doses under 80 mg of APG-1252 will be explored as monotherapy. Maximum tolerated dose (MTD)/RP2D is defined as the highest dose with ≤ 1/6 patients with dose limiting toxicities. A maximum of 6 patients will be treated at the APG-1252 monotherapy dose level to further characterize safety. Part 2 will commence once APG-1252 monotherapy MTD/RP2D is determined following review of safety and tolerability of APG-1252 monotherapy and discussion between sponsor and investigators. In Part 2, APG-1252 will be tested in combination with ruxolitinib. Part 2 will evaluate tolerability and clinical benefit of the combination APG-1252 plus ruxolitinib using a 3+3 dose escalation design. Patients starting APG-1252 treatment as an addition to ruxolitinib should have been on ruxolitinib daily dose for at least 5 days at the same dose. If they were on fedratinib they should discontinue fedratinib and switch to ruxolitinib for at least 5 days before the addition of APG-1252. The starting dose of APG-1252 in Part 2, will be one dose level lower than the MTD of APG-1252 as monotherapy (i.e, at 80 mg if MTD is 160 and 160 mg if MTD is 240 mg) and will be increased to a maximum of 240 mg once per week, added to ruxolitinib. Once the MTD/RP2D of combination arm is determined, additional patients up to a maximum of 15 will be treated at the RP2D to further evaluate safety and clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed myelofibrosis requiring therapy including:

  1. Either primary or post essential thrombocythemia/polycythemia vera
  2. Have intermediate-2 or high-risk myelofibrosis by International Prognostic Scoring System (IPSS) scoring system
  3. If intermediate-1 myelofibrosis must have palpable splenomegaly ≥ 5 cm below left costal margin
  4. Either in chronic (CP) or accelerated phase (AP)
  5. Patients can be either JAK2 wild type or JAK2V617F mutated
* Patients must be ineligible or unwilling to undergo a stem cell transplantation or receive any other approved standard of care at the time of study entry
* Patients have been previously treated with a JAK inhibitor (JAKi) and are intolerant, resistant, refractory or lost response to the JAKi ruxolitinib or fedratinib, or had sub-optimal response to ruxolitinib. Patients in Part 1 will be those ineligible to receive ruxolitinib and other approved standard of care. (Patients will be defined as having received sub-optimal response to ruxolitinib if, they achieved inadequate response to ruxolitinib based therapy after 6 months of treatment, or had been on a stable dose of ruxolitinib based therapy for < 24 weeks and had shown initial response but in opinion of investigators were unlikely to benefit from continuing dose and schedule of ruxolitinib).
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
* Adequate bone marrow function:

  1. Absolute neutrophil count (ANC) ≥ 0.750 X 10˄9/L
  2. Hemoglobin (Hb) ≥ 9.0 g/dL
  3. Platelets count ≥ 50 X 10˄9/L (independent of transfusion within14 days of first dose)
  4. International normalized ratio (INR), prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤1.5 X upper limit of normal (ULN) unless the subject is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Adequate renal and liver function as indicated by:

  1. Direct bilirubin < 2.0 mg/dL (unless Gilbert's syndrome and evidence of hemolysis)
  2. Serum creatinine < 1.5 mg/dL, if >1.5 mg/dL, creatinine clearance must be ≥ 50 mL/min
  3. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (unless considered to be related to myelofibrosis or patient has known history of Gilberts)
  4. Alkaline phosphatase < 2.5 x ULN
  5. Albumin ≥ 2.5g/dl
* Willingness to use contraception method that is deemed effective by the investigator by female patients of child bearing potential (postmenopausal women amenorrhea for at least 12 months to be considered of non-childbearing potential) and males with partners of child bearing potential, throughout the treatment period and for at least three months following the last dose of study drug
* Ability to understand and willingness to sign a written informed consent form
* Willingness and ability to comply with study procedures and follow-up examination

Exclusion Criteria:

* Received standard or experimental therapy within 14 days or 5 half-lives (whichever is greater) before starting study therapy
* Previously received other B-cell lymphoma-extra large (Bcl-xL) inhibitors
* Receiving concomitant anticancer therapy, except hormonal therapy and patients on ruxolitinib
* Disease associated with myelofibrosis such as metastatic carcinoma, lymphoma, myelodysplasia, hairy cell leukemia, mast cell disease or acute leukemia
* Radiation within 14 days of study entry, thoracic radiation within 28 days of study entry
* Has gastrointestinal conditions that could affect the absorption of oral medication
* Has known active central nervous system (CNS) involvements
* Lack of toxicity recovery from previous therapy ≤ grade 1 or baseline (except alopecia, hemoglobin, neutropenia and thrombocytopenia)
* Use of therapeutic anticoagulants
* Failure to recover adequately, as judged by the investigator, from prior surgical procedures. Patients with active wound healing, patients who have had major surgery within 28 days from study entry, and patients who have had minor surgery within 14 days of study entry
* Unstable angina, or other significant cardiac condition including:

  1. Unstable arrhythmia on treatment including permanent cardiac pacemaker
  2. History of symptomatic congestive heart failure (New York Heart Association [NYHA] Class III or IV)
  3. History of myocardial infarction within 6 months of enrollment
  4. Current unstable angina
  5. Family history of long QT syndrome or corrected QT interval (QTc) (Fridericia or Bazett) > 480 msec
* Active infection requiring systemic antibiotic/ antifungal medication, known clinically active hepatitis B or C infection, or on antiretroviral therapy for HIV disease
* Uncontrolled concurrent illness including, but not limited to: psychiatric illness/social situations that would limit compliance with the study requirements or any other condition or circumstance that would, in the opinion of the investigator, make the patient unsuitable for participation in the study
* Women who are pregnant, breast feeding or women of child-bearing potential (WOCBP) not using an effective method of birth control. WOCBP are sexually active mature women who have not undergone a hysterectomy or who have not been achieved post-menopause for at least 12 consecutive months. WOCBP must have a negative serum pregnancy test with 72 hours of receiving the first dose of study medication
* Male patients whose sexual partners are WOCBP not using effective birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rate at each dose level | 28 days
  DLT will be assessed within the first 28-day cycle of study treatment via CTCAE version 5.0
Spleen Volume Measurement Reduction | 24 weeks
  At least a 35% reduction in spleen volume or ≥ 50% reduction in myelofibrosis related total symptom score (TSS)

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Ascentage Pharma Group Inc.
Locations (2):
- United States (2):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No